CLINICAL TRIAL: NCT05716776
Title: Effect of Axial Length on Peripapillary Retinal Nerve Fibre Layer (RNFL) Using Optical Coherence Tomography (OCT)
Brief Title: Effect of Axial Length of the Globe on Retinal Nerve Fibre Thickness
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Asmaa Ibrahim Mostafa, Principal Investigator, ophthalmology resident, Sohag University
Other Study IDs: Soh-Med-22-12-01
Record Dates: First submitted 2023-01-08; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Myopia
Keywords: Axial length; RNFL
MeSH Terms: conditions — Myopia | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1 short axial length (AL): Axial length less than 21
  Interventions: Diagnostic Test: Optical coherence tomography (OCT)
- Group 2 average axial length (AL): Axial length 21-24
  Interventions: Diagnostic Test: Optical coherence tomography (OCT)
- Group 3 long axial length (AL): Axial length more than 24
  Interventions: Diagnostic Test: Optical coherence tomography (OCT)

INTERVENTIONS:
Diagnostic Test: Optical coherence tomography (OCT) — Measurement of retinal nerve fibre layer (RNFL) thickness using optical coherence tomography

SUMMARY:
the goal of this obsrevational study is to learn about retinal nerve fibres and if their numbers changed with axial length of the globe or not. the main question to answer is there is effect of long axial length on the thickness of the retinal nerve fibers participants will be asked to:

* measure the axial length with ultrasound
* measure the thickness of retinal nerve fibers with optical coherence tomography

DETAILED DESCRIPTION:
Aim of the work:

To investigate the effect of axial length on the peripapillary retinal nerve fiber layer.

Patients and methods Study design: Cross sectional comparative study. Location: Ophthalmology department, Sohag teaching hospital. Ethical approval: A written informed consent will be taken from all patients about the aim of the study, the nature of the planned investigation. An approval of the ethical committee of Sohag Faculty of Medicine will be fulfilled.

Methodology The study will include 80 patients healthy volunteers who underwent ophthalmologic examinations including retinal nerve fiber layer (RNFL) thickness analysis with optical coherence tomography (OCT), auto refraction, and axial length measurement.

Inclusion criteria:

Healthy volunteers attending the outpatient clinic for surface ocular diseases.

Exclusion criteria:

* Glaucoma patients.
* Media opacity (corneal, lens or vitreous opacity)
* Previous ocular surgery.
* Diabetic patients.
* Retinal diseases.

Method of the study:

1. Detailed ophthalmological and medical history.
2. Detailed slit lamp examination.
3. Visual acuity (VA) and best corrected visual acuity (BCVA) using Snellen chart and recorded in decimal notation.
4. Auto refraction using Topcon auto refractometer RM-800.
5. Optical coherence tomography (OCT) scan of retinal nerve fiber layer (RNFL) and ganglion cell complex (GCC) thickness using Avanti scanner Optovue.
6. Axial length (AL) measured by E-Z scan 5500 sonomed A-scan ultrasound and biometry.

The patients will be divided into 3 groups:

Group 1 patients with axial length less than 21 mm. Group 2 patients with axial length 21-24 mm. Group 3 patients with axial length more than 24 mm.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers attending the outpatient clinic for surface ocular diseases.
* patients who are cooperative with optical coherence tomography (OCT) device.

Exclusion Criteria:

* Glaucoma patients.
* Media opacity (corneal, lens or vitreous opacity)
* Previous ocular surgery.
* Diabetic patients.
* Retinal diseases.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Outpatient ophthalmology clinic
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Retinal nerve fibre layer (RNFL) thickness | average of one year
  Measuring Retinal nerve fibre layer (RNFL)thickness using OCT

CONTACTS AND LOCATIONS:
Overall Officials: Engy Mo Mostafa, MD, Study Director — Sohag University

IPD SHARING:
Plan to Share IPD: No